CLINICAL TRIAL: NCT02326675
Title: Randomized Controlled, Open-Label Study on the Use of Cryotherapy in the Prevention of Chemotherapy-Induced Mucositis in Stem Cell Transplant Patients
Brief Title: Cryotherapy in the Prevention of Chemotherapy-Induced Mucositis in Stem Cell Transplant
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis: results of the analysis showed no significant difference between the two study groups
Sponsor: University of Florida (Other)
Collaborators: University of Florida Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB201400628
Record Dates: First submitted 2014-12-12; First posted 2014-12-29 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Mucositis; Hematopoietic Stem Cell Transplantation; Peripheral Blood Stem Cell Transplantation; Stomatitis
Keywords: Etoposide; Cryotherapy
MeSH Terms: conditions — Mucositis; Stomatitis | interventions — Ice; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryotherapy Group (Group A) (Active Comparator): Subjects in the intervention group will receive both standard oral care and cryotherapy. During the 30 minute cryotherapy periods, subjects will eat ice chips, and/or consume very cold or frozen foods. Cryotherapy will begin 15 minutes prior to the start time of each etoposide infusion. After 30 minutes of cryotherapy, subjects will begin the saline rinses. The subject should perform 3 saline rinses over 15 minutes. After 15 minutes of saline rinses, the 30-minute cryotherapy / 15-minute saline rinse cycles will be repeated until 30 min after completion of etoposide infusion (approximately 150 minutes). In addition, an oral care diary will be completed by the subject, and a daily oral assessment will be performed by the investigators.
  Interventions: Other: Ice
- Standard Oral Care Group (Group B) (Active Comparator): Subjects in the control group will receive standard oral care only. At the beginning of each etoposide infusion, the subject will begin the saline rinses. The subject will perform 3 saline rinses over 15 minutes followed by 30 minutes of rest (no rinses). The 15-minute saline rinse / 30-minute rest cycles will be repeated until 30 minutes after the completion of the etoposide infusion (approximately 150 minutes). In addition, an oral care diary will be completed by the subject, and a daily oral assessment will be performed by the investigators.
  Interventions: Other: Normal Saline Solution

INTERVENTIONS:
Other: Ice — This group will receive cryotherapy, saline rinses, an oral care diary will be completed by the subject, and a daily oral assessment will be performed by the investigators as part of their participation.
  Other Names: Cryotherapy,Ice Chips
  Arms: Cryotherapy Group (Group A)
Other: Normal Saline Solution — This group will receive saline rinses, an oral care diary will be completed by the subject, and a daily oral assessment will be performed by the investigators as part of their participation.
  Arms: Standard Oral Care Group (Group B)

SUMMARY:
Oral mucositis is a common complication of cancer therapy. Mucositis results from damage to the mucosal epithelium after delivery of chemotherapy or radiation treatments designed to treat the cancer. A number of treatment factors have been shown to influence the incidence and severity of mucositis, including chemotherapy type and dosage. High-dose chemotherapy before stem cell transplantation can cause severe oral mucositis and is often the side effect that patients find the most difficult to endure. Cryotherapy, keeping ice chips in the mouth during chemotherapy infusion, has been shown to prevent or alleviate mucositis caused by high-dose melphalan alone or given in combinations used in pre-transplant conditioning. One other drug notorious for causing severe mucositis is etoposide (VP-16). The specific aims of the study are: 1) to assess tolerability of cryotherapy given during chemotherapy administration; 2) to determine the efficacy of cryotherapy in reducing etoposide-induced mucositis.

DETAILED DESCRIPTION:
As a participant the following will happen:

There will be a random assignment (much like the flip of a coin) to one of two study groups:

* Group A: Standard mouth care plus cryotherapy, or
* Group B: Standard mouth care.

Standard Mouth Care plus Cryotherapy (Group A)

Will receive the standard mouth care plus Cryotherapy and will consist of:

* Mouth care 3 times daily with a soft-bristle toothbrush or foam toothbrush
* Cryotherapy - beginning 15 minutes before etoposide chemotherapy starts, the consumption of ice chips and/or other very cold and frozen foods (popsicles, Italian Ice etc.) continuously for 30 minutes.

  o Short (1 to 3 minutes maximum) breaks over the course of the 30 minute period as long as at least 15 minutes are spent actively engaged in the cryotherapy
* Saline "swish and spit" mouth rinses - you will be asked to rinse your mouth with saline for approximately 30 seconds before spitting out the saline into the sink or basin

  o You will be asked to do this 3 times over 15 minutes following each 30 minute period of cryotherapy
* The cycle of 30 minutes of cryotherapy followed by 15 minutes of saline mouth rinses will be repeated until 30 minutes after the etoposide infusion (approximately 3 cycles for a typical 120 minute infusion).

Standard Mouth Care (Group B)

Randomization to the Standard Mouth Care group will consist of:

* Mouth care 3 times daily with a soft-bristle toothbrush or foam toothbrush
* Saline "swish and spit" mouth rinse - rinse the mouth with saline for approximately 30 seconds before spitting out the saline into the sink or basin

  * At the beginning of each etoposide infusion, perform three 30-second saline rinses over 15 minutes followed by a 30-minute break from the rinses
  * The cycle of 15-minute saline mouth rinses followed by 30-minute break periods will be repeated until 30 minutes after the etoposide infusion (approximately 3 cycles for a typical 120 minute infusion).

The standard mouth care group, will not be permitted to eat ice chips or consume frozen foods during the times these times.

All groups will have the following interventions and assessments performed:

* Mouth Care Diary - the time and type of mouth care and/or cryotherapy
* Mucositis Assessments - pain levels, appetite, ability to swallow liquids and/or food

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 18 year old or older who are eligible candidates for myeloablative autologous stem cell transplantation (ASCT).
* Subjects receiving etoposide as part of their conditioning regimen with a planned total dose of ≥ 30 mg/kg.

Exclusion Criteria:

* Subjects with prior radiation to head & neck region.
* Subjects with known oropharynx involvement with their malignancy.
* Subjects with a history of non-compliance or who lack capacity to give informed consent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Number of participants that tolerate cryotherapy during each etoposide infusion | Up to seven days prior to stem cell transplant.
Time to onset, severity and duration of mucositis following etoposide administration | Participants will be followed starting on Day +1 post-transplant until they are discharged from the hospital, an expected average of 3-4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Dees, RN, Principal Investigator — UF Health
Locations (1):
- UF Health Shands Cancer Hopsital, Gainesville, Florida, United States